CLINICAL TRIAL: NCT07318064
Title: Ultra-processed Food Consumption and Health Pilot Study
Acronym: ULTRA PIlot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Peter T. Katzmarzyk, Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025-063
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight
Keywords: ultra-processed diet; precision nutrition; metabolomics; weight loss
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Purple Diet (Active Comparator): The Purple Diet is modeled after a typical American diet which is popular, widely available, and lower in cost compared to other diets. However, the diet is high in total fat, and particularly in saturated fat, with consumption far exceeding 10% of total energy intake. Intake of added sugars also far exceeds the recommended limits. The Purple Diet has been used in the Nutrition for Precision Health study.
  Interventions: Behavioral: Purple Diet
- Ultra-processed Diet (Experimental): The ultra-processed (UPF) diet is designed to contain approximately 75% of energy from ultra-processed foods. Foods and ingredients in the ultra-processed diet consist of those defined in the NOVA classification as "ultra-processed" (group 4 of the classification). The NOVA classification groups foods according to the nature, extent and purpose of the industrial processing they undergo.10 In the NOVA classification, ultra-processed foods include such things as soft drinks, packaged snacks, reconstituted meat products and pre-prepared frozen dishes, and are made mostly or entirely from substances derived from foods and additives, with little if any unprocessed foods.
  Interventions: Behavioral: Ultra-processed diet

INTERVENTIONS:
Behavioral: Purple Diet — The Purple Diet is modeled after a typical American diet which is popular, widely available, and lower in cost compared to other diets. However, the diet is high in total fat, and particularly in saturated fat, with consumption far exceeding 10% of total energy intake. Intake of added sugars also far exceeds the recommended limits.
  Arms: Purple Diet
Behavioral: Ultra-processed diet — The ultra-processed food (UPF) diet is designed to contain approximately 75% of energy from ultra-processed foods. Foods and ingredients in the ultra-processed diet consist of those defined in the NOVA classification as "ultra-processed" (group 4 of the classification). The NOVA classification groups foods according to the nature, extent and purpose of the industrial processing they undergo.10 In the NOVA classification, ultra-processed foods include such things as soft drinks, packaged snacks, reconstituted meat products and pre-prepared frozen dishes, and are made mostly or entirely from substances derived from foods and additives, with little if any unprocessed foods.
  Arms: Ultra-processed Diet

SUMMARY:
The objective of this study is to explore the effects of two dietary conditions (UPF-diet and typical American diet) on a number of clinical and metabolic outcomes in order to derive sample size estimates for a larger trial and to determine the feasibility of the study approach.

This study is an out-patient cross-over trial comparing the Nutrition for Precision Health (NPH) purple diet (American Diet) and a diet high in ultra-processed foods (UPF diet) for two weeks in which participants will be randomized to the order of the diets.

Specific Aim 1: Determine the feasibility of recruiting, enrolling and assessing participants in a randomized trial comparing a UPF diet with the standard American diet. Feasibility will be assessed by the achievement of study goals (i.e., sample size; completeness of study data).

Specific Aim 2: Derive sample size estimates for future trials based on the mean effects and associated variances obtained in the pilot study.

DETAILED DESCRIPTION:
The investigators will conduct an out-patient cross-over trial comparing the Nutrition for Precision Health (NPH) purple diet and a diet high in ultra-processed foods (UPF diet) with participants randomized equally to one of two conditions. Assessments of study outcomes will be conducted at baseline prior to randomization, and pre- and post- each dietary condition. The overarching aim is to determine the feasibility of the study approach, and to explore the effects of the dietary conditions on a number of clinical and metabolic outcomes.

Participants in this study will be 6 adults (both males and females) recruited from the community. Participants will receive each dietary condition for 14 days, with at least a 14-day wash-out period between conditions. The order of the conditions will be randomized.

Participants in both intervention conditions will be provided with meals and snacks prepared by the Pennington Biomedical Metabolic Kitchen. The total daily kilocalories, energy density, and macronutrient content of the two diets presented to the participants will be equivalent across the two conditions. Participants will be asked to consume only the foods provided according to a daily menu (including up to 2 cups of coffee or tea), water, and up to 12 oz. of artificially-sweetened beverages, and to adhere to their other usual routines (e.g., exercise, sleep, medication use) throughout the study.

Both diets will be isocaloric and will be provided using 3-day cycle menus, prepared by the Metabolic Kitchen. Menus will provide 3 meals and at least one snack. Participants will have some flexibility to distribute their meals and snacks across each day according to their preference. For menu planning, a 2100 kcal/d diet with scaled adjustments for individual energy needs will be planned. Templates will be developed that consist of 1600kcal, 2100kcal, 2600kcal, 3200kcal, and 3700kcal menus; 100 or 200 kcal foods that conform to the diet pattern and macronutrient profile will be added to the menu template (1600, 2100, 2600, 3200, or 3700 kcal) to deliver energy to the nearest hundred-kcal of estimated energy needs. These foods will also be added or removed from menus in cases of sustained weight loss or weight gain.

Participants will pick up study meals two to three times per week and will be provided with a 2 to 4-day meal supply at each pick-up. Meals will be assembled in advance of participant pick up and according to dietary intervention assignment, energy requirements and the allowed substitutions for food preferences. At the time of food dispensing, the participant's identity will be verified to match the provided meals. Meals will be packaged in a cooler for temperature-controlled transport along with instructions for retherming as needed.

The study outcomes will be collected immediately prior to and after each dietary condition.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity (BMI 25-50 kg/m2)
* Willingness to accept group assignment and provide outcome measures
* Premenopausal (women only)
* Be able to communicate (oral and written) in English
* Be able to provide informed consent

Exclusion Criteria:

* Recent weight loss (≥10 pounds in the last six months)
* On a regimen of medications (weight loss or otherwise) that can affect weight or diabetes outcomes for less than 3 months (GLP1 medications allowed if weight stable and on stable dose for >=3 months)
* Given birth within the past year or is currently pregnant or breastfeeding
* Past bariatric surgery (<10 years) - all types
* Disease/condition that is life threatening or can interfere with or be aggravated by weight change
* Dementia, psychiatric illness, or substance abuse that may interfere with adherence
* Current or history of a clinically diagnosed eating disorder, including anorexia nervosa or bulimia nervosa
* Type 1 or type 2 diabetes
* Uncontrolled gastrointestinal disorders including chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, chronic diarrhea or active gallbladder disease
* Current cancer or cancer treatment, or a history of cancer or cancer treatment within the last 3 years. Exceptions include 1) successfully resected non-melanoma carcinoma of the skin, 2) basal or squamous cell skin cancer, 3) stage 0 non-invasive carcinoma of the cervix, 4) stage 0 non-invasive prostate cancer
* History of kidney or liver disease or malnutrition that in investigator judgment should exclude participation
* Hemoglobinopathy that interferes with measurement of HbA1c
* Class II or higher congestive heart failure
* Unstable heart disease
* Blood pressure ≥160/100 mm Hg
* Thyroid disease for which the participant is untreated or has had treatment changed within the last 6 weeks.
* Unwilling to stop alcohol intake during study participation
* Current smoker or other type of tobacco user (chewing tobacco, vaping, etc.)
* Any other condition or factor which in the opinion of the study physician or investigator makes it inadvisable for the candidate to participate in the trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Body weight | Change from baseline to 14 days
  Body weight measured in kg

SECONDARY OUTCOMES:
Physical activity | Change from baseline to 14 days
  Physical activity measured using the International Physical Activity Questionnaire - Short Form (IPAQ-SF)
Waist circumference | Change from baseline to 14 days
  Waist circumference measured in cm
Total body fat | Changes from baseline to 14 days
  Total body fat in kg measured using Dual-Energy X-Ray Absorptiometry (DXA)
Total fat-free mass | Change from baseline to 14 days
  Fat free mass in kg measured using Dual-Energy X-ray Absorptiometry (DXA)
Twenty-four-hour interstitial glucose | Continuously from baseline to 14 days
  Twenty-four-hour interstitial glucose will be measured using continuous glucose monitoring
Systolic blood pressure | Change from baseline to 14 days
  Resting systolic blood pressure will be measured in mmHg
Diastolic blood pressure | Change from baseline to 14 days
  Resting diastolic blood pressure measured in mmHg
Total cholesterol | Change from baseline to 14 days
  Total cholesterol measured in mg/dL
Triglycerides | Change from baseline to 14 days
  Triglycerides measured in mg/dL
HDL-cholesterol | Change from baseline to 14 days
  HDL-cholesterol measured in mg/dL
LDL-cholesterol | Change from baseline to 14 days
  LDL-cholesterol measured in mg/dL
Glucose | Change from baseline to 14 days
  Fasting glucose measured in mg/dL
Insulin | Change from baseline to 14 days
  Fasting insulin measured in mg/dL
HbA1c | Change from baseline to 14 days
  HbA1c measured in %
Appetite | Change from baseline to 14 days
  Appetite ratings (hunger/fullness/desire to eat) will be measured using visual analog scales.
Cognitive restraint | Change from baseline to 14 days
  Cognitive restraint will be measured using the three-factor eating Questionnaire (TFEQ)
Disinhibition | Change from baseline to 14 days
  Disinhibition will be measured using the Three-Factor Eating Questionnaire (TFEQ)
Hunger | Change from baseline to 14 days
  Hunger will be measured using the Three-Factor Eating Questionnaire (TFEQ)

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Katzmarzyk, PhD, Principal Investigator — Pennington Biomedical Research Center

IPD SHARING:
Plan to Share IPD: Yes
Raw deidentified data on the primary and secondary outcome measures collected during the trial will be available.
Supporting Information: Study Protocol
Time Frame: Data will be available indefinitely starting from the publication of the primary paper.
Access Criteria: Data will be stored in the Pennington Biomedical Nutrition Obesity Research Center (NORC) Data and Biorepository. Data are available upon reasonable request to the repository manager.